CLINICAL TRIAL: NCT06322758
Title: Driving Pressure-guided Tidal Volume Ventilation in the Acute Respiratory Distress Syndrome: a Prospective, Multicenter, Randomized, Controlled, Open-label, Phase III Trial
Brief Title: Driving Pressure-guided Tidal Volume Ventilation in the Acute Respiratory Distress Syndrome
Acronym: DRIVENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230851
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Distress Syndrome ARDS
Keywords: Acute respiratory distress syndrome (ARDS); ventilator-induced lung injury (VILI); respiratory system compliance (Crs); tidal volume (VT); driving pressure (ΔP); predicted body weight (PBW)
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury; Acrocephalosyndactylia

STUDY DESIGN:
Intervention Model Description: comparing ΔP-guided VT to traditional PBW-guided VT during mechanical ventilation of patients with ARDS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ΔP-guided VT group (Experimental): During volume assist control ventilation, the VT will be adjusted in supine position to target a 12 ≤ ΔP ≤ 14 cm H2O. The allowed minimal and maximal values of VT are consistent with usual practices reported in large observational studies 4 and 10 mL/kg of PBW, respectively, while keeping a plateau pressure below 30 cm H2O. The respiratory rate will then be adjusted to meet the pH target
  Interventions: Other: Tidal volume customization in the acute respiratory distress syndrome
- PBW-guided VT group (Active Comparator): The VT will be kept at 6 mL/kg of PBW. If the plateau pressure threshold is reached (30 cm H2O), the VT will be decreased down to a minimal value of 4 mL/kg of PBW.
  Interventions: Other: Tidal volume customization in the acute respiratory distress syndrome

INTERVENTIONS:
Other: Tidal volume customization in the acute respiratory distress syndrome — During volume assist control ventilation, the VT will be adjusted in supine position to target a 12 ≤ ΔP ≤ 14 cm H2O. The allowed minimal and maximal values of VT are consistent with usual practices reported in large observational studies 4 and 10 mL/kg of PBW, respectively, while keeping a plateau pressure below 30 cm H2O. The respiratory rate will then be adjusted to meet the pH target

SUMMARY:
Acute respiratory distress syndrome (ARDS) is associated with high mortality, some of which can be attributed to ventilator-induced lung injury (VILI) when artificial ventilation is not customized to the severity of lung injury. As ARDS is characterized by a decrease in aerated lung volume, reducing tidal volume (VT) from 12 to 6 mL/kg of predicted body weight (PBW) was shown to improve survival more than 20 years ago. Since then, the VT has been normalized to the PBW, meaning to the theoretical lung size (before the disease), rather than tailored to the severity of lung injury, i.e., to the size of aerated lung volume. During ARDS, the aerated lung volume is correlated to the respiratory system compliance (Crs). The driving pressure (ΔP), defined as the difference between the plateau pressure and the positive end expiratory pressure, represents the ratio between the VT and the Crs. Therefore, the ΔP normalizes the VT to a surrogate of the aerated lung available for ventilation of the diseased lung, rather than to the theoretical lung size of the healthy lung, and thus represents more accurately the actual strain applied to the lungs. In a post hoc analysis of 9 randomized controlled trials, Amato et al. found that higher ΔP was a better predictor of mortality than higher VT, with an increased risk of death when the ΔP > 14 cm H2O. These findings have been confirmed in subsequent meta-analysis and large-scale observational data. In a prospective study including 50 patients, the investigators showed that a ΔPguided ventilation strategy targeting a ΔP between 12 and 14 cm H2O significantly reduced the mechanical power, a surrogate for the risk of VILI, compared to a conventional PBW-guided ventilation. In the present study, the investigators hypothesize that the physiological individualization of ventilation (ΔP-guided VT) may improve the outcome of patients with ARDS compared to traditional anthropometrical adjustment (PBW-guided VT)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Invasive mechanical ventilation
* Criteria for ARDS according to Berlin definition:
* Bilateral infiltrates not fully explained by effusions, lobar/lung collapse, or nodules;
* PaO2/FiO2 of 300 or less measured with a PEEP of at least 5 cm H2O
* Respiratory failure not fully explained by cardiac failure or fluid overload These criteria must be observed for less than 72h
* Affiliation to the social security system
* Written consent obtained from the patients (from a support person, family member or a close relative if the patient is not able to expressing and sign consent) or inclusion without initial consent in case of emergency, if the patient is not able to express his/her consent and in the absence of support person, family member or a close relative

Exclusion Criteria:

* Known pregnancy
* Lung transplantation
* Evident significant decrease in chest wall compliance (e.g., abdominal compartment syndrome)
* Moribund patient not expected to survive 24 hours
* Presence of an advanced directive to withhold life-sustaining treatment or decision to withhold life-sustaining treatment
* Chronic respiratory disease requiring home oxygen therapy or ventilation
* ECMO before inclusion
* Pneumothorax
* Enrollment in an interventional ARDS trial with direct impact on VT
* Subject deprived of freedom, subject under a legal protective measure (guardianship/curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  The primary endpoint is a ranked composite score that prioritizes 28-day mortality, followed by days free from mechanical ventilation through day 28 for the survivors. Thus, the score is calculated in such a manner that death constitutes a worse outcome than fewer days off the ventilator.
Number of days free from mechanical ventilation | 28 days
  The primary endpoint is a ranked composite score that prioritizes 28-day mortality, followed by days free from mechanical ventilation through day 28 for the survivors. Thus, the score is calculated in such a manner that death constitutes a worse outcome than fewer days off the ventilator.

SECONDARY OUTCOMES:
Ventilator parameters | up to Day 7
Arterial blood gases | up to Day 7
  Arterial blood gases (pH, PaO2, PaCO2, HCO3-), recorded in supine position between 6:00 and 12:00 a.m. once a day up to day 7
Mortality | Day-28, Day 90
  ICU mortality and hospital mortality
Number of days alive without ventilation | Up to Day 28
  Number of days alive without ventilation between randomization and day 28;
Sequential Organ Failure Assessment score (SOFA) | Day 1, Day 3 and Day 7
  SOFA score
Number of days alive without catecholamine | Up to Day 28
  Number of days alive without catecholamine between randomization and day 28, assessed as a hierarchical endpoint prioritized on 28-day mortality;
Number of days alive without continuous sedation | Up to Day 28
  Number of days alive without continuous sedation between randomization and day 28, assessed as a hierarchical endpoint prioritized on 28-day mortality
Number of days alive without neuromuscular blockers | UP to Day 28
  Number of days alive without neuromuscular blockers between randomization and day 28, assessed as a hierarchical endpoint prioritized on 28-day mortality;
Number of prone position sessions | Up to Day 28
  Number of prone position sessions
Use of rescue procedures: inhaled nitric oxide, almitrine, ECMO, ECCO2R | Up to Day 28
  Use of rescue procedures: inhaled nitric oxide, almitrine, ECMO, ECCO2R
Occurrence of ventilator-associated pneumothorax | Up to Day 28
  Occurrence of ventilator-associated pneumothorax between randomization and day 28;
Time to pressure support ventilation; | Up to Day 28
  Time between randomization and transition to pressure support ventilation;
Duration of weaning unreadiness | Up to Day 28
  Duration of weaning unreadiness measured as the time between randomization and initiation of weaning from mechanical ventilation, defined as the day of the first spontaneous breathing trial;
Duration of weaning | Up to day 28
  Duration of weaning, defined as the time between the first spontaneous breathing trial and successful extubation
The rate of tracheostomy | Up to Day 28
  The rate of tracheostomy
Total duration of mechanical ventilation | up to Day 7
  Total duration of mechanical ventilation, from intubation to successful extubation, defined as an extubation not followed by reintubation or death within the next 7 days;
Length of stay | up to Day 28
  Length of stay in the ICU and in hospital;

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION